CLINICAL TRIAL: NCT02905903
Title: An In Vivo Model for Postinflammatory Hyperpigmentation: Part II
Brief Title: An In Vivo Model for Postinflammatory Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB #9920 Protocol 1
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Post-inflammatory Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trichloroacetic Acid (Other): Intervention-Apply 4 concentrations of TCA (20%, 25%, 30%, 35%) to the buttocks to two spots each (total of 8 lesions) and following characteristics of these lesions and comparing them to acne induced PIH during the course of the study. Comparisons will be made using Investigators Global Assessment scoring of hyperpigmentation and erythema, colorimetry, photography, and biopsies
  Interventions: Drug: Tricholoacetic Acid (TCA)

INTERVENTIONS:
Drug: Tricholoacetic Acid (TCA) — We will be applying 4 concentrations of TCA (20%, 25%, 30%, 35%) to the buttocks to two spots each (total of 8 lesions) and following characteristics of these lesions and comparing them to acne induced PIH during the course of the study.

SUMMARY:
Post-inflammatory hyperpigmentation (PIH) is an acquired hypermelanosis that occurs after cutaneous inflammation or injury that frequently affects darker skinned populations. Previously, a model of 35% TCA-induced PIH was validated against acne induced PIH, which has value in product testing for the treatment of PIH. In this second phase of the study, the investigators would like to determine if a lower concentration of TCA-induced PIH is comparable to acne-induced PIH.

DETAILED DESCRIPTION:
Post-inflammatory hyperpigmentation (PIH) is an acquired hypermelanosis that occurs after cutaneous inflammation or injury. This process can occur in all skin types but more frequently affects darker skinned patients, such as African-Americans, Hispanics, Asians, Native Americans, Pacific Islanders and those of Middle Eastern descent. PIH can occur after infection, allergic reactions, contact dermatitis, some medications, burns, following procedures, or inflammatory disease such as acne. In skin of color, PIH frequently occurs in resolving acne lesions and can persist for months after the acne lesion itself has disappeared. In many cases, the resulting PIH can be more distressing than the original insult.

During the first phase of this study, the investigators investigated the clinical, spectroscopic and histologic characteristics of acne-induced PIH versus irritant induced PIH using Trichloroacetic acid (TCA), 35% solution. From this initial study, the investigators concluded that the similarity of Investigator's Global Assessment scores, and spectroscopic measurements using Diffuse Reflectance Spectroscopy and Colorimetry in both acne and TCA-induced PIH at Day 28 suggest that TCA-induced PIH could be a reproducible model for acne induced PIH.

MicroRNAs (miRNAs) are a class of small non-coding RNA molecules that regulate the expression of multiple genes at the post-transcriptional level through degradation and translation of target mRNAs. In the initial study, the investigators hypothesized that miRNAs derived from melanocytes and immune cells during PIH development could be detected in tissue and serve as novel biomarkers for PIH and making appropriate therapeutic decisions. To test this hypothesis, the investigators first examined miRNA gene expression profiles during PIH development using different models, and then evaluated miRNAs profiles in acne- induced PIH, TCA- induced PIH and normal skin. The investigators have defined some miRNAs that potentially are involved in PIH development and may be also serve as the biomarkers for PIH. The investigators found that there were 19 miRNA changes in acne-induced PIH versus normal skin, while 43 miRNA changes in TCA-inducedPIH versus normal skin. Interestingly, about 80% changed genes in acne were included in TCA-mediated miRNA changes, suggesting TCA can partially mimic acne-PIH.

Overall, this initial model for PIH, using TCA, serves as a foundation to better understand and improve our ability to manage PIH. In this next phase of the study, the investigators will refine this in vivo model for PIH by determining the optimal concentration of TCA to induce PIH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with types I-VI skin
* Minimum age of 18 years
* Able to understand requirements of the study and risks involved
* Able to sign a consent form.
* Existing truncal acne pustules (at least two on the trunk) with or without history of post-inflammatory hyperpigmentation

Exclusion Criteria:

* Patients with a recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of PIH judged to be clinically significant by the investigator
* Patients with a history of keloids
* Patients with a history of cystic acne or acne conglobata
* Patients on systemic antibiotics or keratolytics (isotretinoin, etc), or topical antibiotics or keratolytic use (retinoids, benzoyl peroxide) over target areas who are unwilling to stop these medications for the duration of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-14 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Optimal TCA concentration for induction of post-inflammatory hyperpigmentation | 35 days
  This will be determined by comparing acne induced PIH and the different concentrations of TCA induced PIH
Study genetic components of post-inflammatory hyperpigmentation by evaluating single nucleotide polymorphism and microRNA | 35 days
  These will be evaluated by blood draws and biopsy
Study individual risk factors for those susceptible to developing postinflammatory hyperpigmention | 35 days
  These will be evaluated by surveys and comparing subjects with PIH versus no PIH

SECONDARY OUTCOMES:
validate a quality of life questionnaire for post-inflammatory hyperpigmentation. | 35 days
  Administration of PIH surveys

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor S, Grimes P, Lim J, Im S, Lui H. Postinflammatory hyperpigmentation. J Cutan Med Surg. 2009 Jul-Aug;13(4):183-91. doi: 10.2310/7750.2009.08077. PMID 19706225
- [Background] Davis EC, Callender VD. Postinflammatory hyperpigmentation: a review of the epidemiology, clinical features, and treatment options in skin of color. J Clin Aesthet Dermatol. 2010 Jul;3(7):20-31. PMID 20725554
- [Background] Baumann L, Rodriguez D, Taylor SC, Wu J. Natural considerations for skin of color. Cutis. 2006 Dec;78(6 Suppl):2-19. PMID 17354519
- [Background] Grimes PE, Stockton T. Pigmentary disorders in blacks. Dermatol Clin. 1988 Apr;6(2):271-81. PMID 3378372
- [Background] Motokawa T, Kato T, Hashimoto Y, Katagiri T. Effect of Val92Met and Arg163Gln variants of the MC1R gene on freckles and solar lentigines in Japanese. Pigment Cell Res. 2007 Apr;20(2):140-3. doi: 10.1111/j.1600-0749.2007.00364.x. PMID 17371441
- [Background] Szell M, Baltas E, Bodai L, Bata-Csorgo Z, Nagy N, Dallos A, Pourfarzi R, Simics E, Kondorosi I, Szalai Z, Toth GK, Hunyadi J, Dobozy A, Kemeny L. The Arg160Trp allele of melanocortin-1 receptor gene might protect against vitiligo. Photochem Photobiol. 2008 May-Jun;84(3):565-71. doi: 10.1111/j.1751-1097.2008.00296.x. Epub 2008 Feb 11. PMID 18282185